CLINICAL TRIAL: NCT00287937
Title: Phase I Study Of Suberoylanilide Hydroxamic Acid (SAHA) (NSC 701852) in Combination With Paclitaxel /Carboplatin for Advanced and Refractory Solid Malignancies
Brief Title: Vorinostat, Paclitaxel, and Carboplatin in Treating Patients With Advanced or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02676; PHI 51; U01CA099168 (NIH); U01CA062505 (NIH); CDR0000454713 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Vorinostat; Paclitaxel; Taxes; Carboplatin

ARMS (1):
- Treatment (vorinostat, paclitaxel, carboplatin) (Experimental): Patients receive oral SAHA once or twice daily on days 1-14* and paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who have stable disease after the completion of 6 courses may receive single-agent SAHA at the discretion of the treating physician.
  Interventions: Drug: vorinostat; Drug: paclitaxel; Drug: carboplatin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with paclitaxel and carboplatin in treating patients with advanced or refractory solid tumors. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with paclitaxel and carboplatin may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the recommended phase II dose of vorinostat (SAHA) when administered with paclitaxel and carboplatin in patients with advanced or refractory solid tumors.

SECONDARY OBJECTIVES:

I. Determine the dose-limiting toxicity (DLT) and other toxic effects of this regimen in these patients.

II. Assess, preliminarily, evidence of antitumor activity of this regimen in these patients.

III. Determine the pharmacokinetic parameters of this regimen in these patients.

IV. Determine the in vivo effects of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of vorinostat (SAHA).

Patients receive oral SAHA once or twice daily on days 1-14* and paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who have stable disease after the completion of 6 courses may receive single-agent SAHA at the discretion of the treating physician.

NOTE: *During the first treatment course only, patients receive SAHA on days -4 to 10.Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT. An additional 6-12 patients are treated at the MTD.

After completion of study treatment, patients are followed at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor
* No untreated brain metastases

  * Patients with stable brain disease (no concurrent corticosteroids) ≥ 4 weeks after completion of appropriate therapy are eligible
* ECOG performance status ≤ 2 OR Karnofsky performance status 60-100%
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double barrier contraception for at least 1 week before, during, and for at least 2 weeks after study participation
* No peripheral neuropathy > grade 1
* No history of allergic reactions to paclitaxel
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs
* No inability to take oral medications on a continuous basis
* No psychiatric illness or social situation that would limit compliance with this study
* No ongoing or active infection
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No other uncontrolled illness
* No more than 2 prior chemotherapy regimens for advanced/metastatic disease

  * Adjuvant chemotherapy administered ≥ 2 years prior to study entry is not considered a prior chemotherapy regimen for purposes of this study
* No prior therapy with paclitaxel
* No chemotherapy or radiotherapy within the past 3 weeks (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 4 weeks since prior valproic acid
* No other concurrent anticancer therapies or agents
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent oral contraceptives
* No concurrent prophylactic growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-07; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
MTD of vorinostat defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT | 21 days

SECONDARY OUTCOMES:
Toxicity graded using the CTC version 2.0 | Up to 1 month after completion of study treatment
  Tables will be created to summarize these toxicities by dose and by course.
Overall survival | Up to 1 month after completion of study treatment
  Summarized with Kaplan-Meier plots.
Time to failure | Up to 1 month after completion of study treatment
  Summarized with Kaplan-Meier plots.
Response defined using the RECIST criteria | Up to 1 month after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States